CLINICAL TRIAL: NCT06219122
Title: The Effectiveness of a Creative Arts en Psychomotor Therapy Intervention for People With Personality Disorders to Enhance Psychological Adaptation and Wellbeing, a Multiple Baseline Single Case Experimental Design.
Brief Title: The Effectiveness of a Creative Arts en Psychomotor Therapy Intervention for People With Personality Disorders. From Negative Thinking to Positive Acting.
Acronym: NDPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzanne Haeyen (Other)
Collaborators: University of Twente (Other)
Responsible Party: Sponsor-Investigator, Suzanne Haeyen, dr. Suzanne Haeyen, professor of arts and psychomotor therapies, HAN University of Applied Sciences
Organization: HAN University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NDPD - SU1606
Record Dates: First submitted 2023-12-22; First posted 2024-01-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Personality Disorders
Keywords: Personality Disorders; Mental wellbeing; Creative arts and Psychomotor therapies
MeSH Terms: conditions — Personality Disorders

STUDY DESIGN:
Intervention Model Description: Multiple baseline single case experimental design wherein all patients are first assigned to the control condition (or control period) and are then assigned to the intervention condition (or intervention period) and finally the follow-up period (control period). Patients are randomized for the time (t) at which they start with the intervention. CONSORT recognizes this design as an N=1 Trial, please refer to https://www.consort-statement.org/extensions/overview/n-of-1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A CAPTS intervention for people with personality disorders. (Experimental): Experimental: Control Period - Intervention Period Multiple baseline single case experimental design wherein all patients are first assigned to the control condition (or control period) are then assigned to the intervention condition (or intervention period) and finally to the follow-up period (control period). Patients are randomized for the time (t) at which they start with the intervention.
  Interventions: Behavioral: Creative arts and psychomotor therapies intervention for people with personality disorders

INTERVENTIONS:
Behavioral: Creative arts and psychomotor therapies intervention for people with personality disorders — a Group (max of 9 participants) Creative arts and psychomotor therapies (CAPTS) intervention for people with personality disorders. Consisting of 10 sessions, where two CAPTS disciplines and therapists are represented each session. Each session lasts 90 minutes. Sessions are aimed at psychological adativity thru=ough the CAPTS. The sessions cover warming up in one of the CAPTS, short psycho education and a longer assigment focusing on the session goal. The first half of the interventions focusses mainly on listening to body signals, emotions and emotional needs and dealing in a healthy way with these. The second half will be more complex when dealing with challenges and adapting tot he context in a healthy way are goals of the sessions.

SUMMARY:
Mental health consists of the absence of mental disorders and the presence of mental well-being. However; mental health care currently focuses mainly on mental disorders and less on promoting mental well-being. And yet people with personality problems often score very low on well-being. In order to work on sustainable mental health, attention is needed for both mental complaints and well-being and this is achieved through promoting psychological adaptation.

Psychological adaptation is the process in which a person deals in a healthy way with their own needs, emotions and inner signals (such as stress) as well as the smaller or larger challenges in life. For people with personality problems psychological adaptation is also low, they mainly react in rigid patterns.

Creative arts and psychomotor therapies (CAPTS) are a non-verbal form of therapy in which various creative methods, such as theater, sports, dance, music and sports methods, are used to make contact with emotions and to practice healthier ways of dealing with them. This is very suitable for working on promoting psychological adaptivity, within a safe and playful context. It's about doing and experiencing, and discovering what works for you personally, more than talking and understanding.

That this is effective is endorsed by professionals and clients in mental health care, but scientific evidence is still scarce. That is why a specially developed, CAPTS module for people with personality problems will be investigated in a mixed methods design. We focus on both effectiveness and working mechanisms in a Multiple Baseline Single Case Experimental Design and a qualitative approach.

DETAILED DESCRIPTION:
Personality disorders are common psychiatric disorders. 5%-10% of all Dutch people have a personality disorder. The best-known personality disorders are borderline, narcissistic and avoidant personality disorders. Personality disorders often arise in adolescence. Deep-seated limitations in behavior, thoughts, feelings, connection and intimacy lead to long-term dysregulation in dealing with oneself and others. This causes problems in several areas of life that patients can no longer solve themselves, including difficulties in intimate relationships and incapacity for work. Specialist treatment can turn the tide.

Creative arts and psychomotor therapies (CAPTS) are often a permanent part of the treatment for personality disorders, in addition to psychotherapy and psychotropic drugs. The treatment tradition of the CAPTS spans approximately a century and includes the disciplines: art, drama, dance, music and psychomotor therapy. For professional therapists, the patients' request for help is the starting point. The treatments for the various personality disorders therefore often overlap. The CAPTS focus on experiencing and doing. Feelings, thoughts and behavioral patterns emerge through making art, play, music or physical sensation. Awareness and (self) reflection are stimulated and new roles and skills are practiced in a safe manner.

With CAPTS, patients with a personality disorder can develop more appropriate ways of relating to themselves and others. To date, little practice-oriented research has been conducted into the treatment of personality disorders with occupational therapy. However, the Dutch Healthcare Institute insists on substantiation of the effectiveness of the CAPTS to justify its reimbursement. There is also an increasing demand for this from the professional organizations of professional therapists and patient organizations.

Existing treatments for personality disorders are aimed at reducing complaints. However, mental health also consists of the presence of well-being. Well-being is about whether someone feels good psychologically, emotionally and socially. Even if patients have physical and psychological complaints. Patients with a personality disorder often have low well-being. Promoting well-being is an important step towards their recovery, which is an important treatment goal according to the treatment guideline. Working on better psychological adaptation is how this can be achieved, one will get more adaptive to their own emotional needs within the context of daily life. Wellbeing will be improved accordingly.

CAPTS professionals indicate that no specific treatment module with CAPTS interventions has yet been developed to promote the psychological adaptation and well-being of patients with a personality disorder. From a professional point of view, they feel the need for this, because that is precisely where their strength lies. Patient organizations confirm the importance of this from the patient perspective.

When developing and evaluating CAPTS interventions, it is therefore important to promote psychological adaptation and well-being of patients with a personality disorder, in addition to reducing complaints.

In summary, personality disorders are common and serious psychiatric disorders that impair psychological and social functioning. CAPTS treatment is promising for promoting psychological adaptation and well-being of patients with personality disorders. However, treatment specifically aimed at this is not yet available in practice. Practical research into the development and evaluation of CAPTS interventions meets an important and immediate need in the professional field and is in line with the treatment guidelines for personality disorders and various national research agendas. From a social perspective, the proper treatment of people with serious psychological suffering is an important issue.

Research Question:

How can the various CAPTS disciplines promote psychological adaptivity in patients with a personality disorder and what is the effect of this approach on complaint reduction and well-being?

Aim of this research:

Designing and testing a practical and broadly applicable module with CAPTS interventions and a practical manual that promote psychological adaptation and well-being of people with personality disorders.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with one or more PD according to the DSM-V criteria
* being motivated for CAPTs
* able to participate in group therapy

Exclusion Criteria:

* acute psychosis or crisis
* prominent PTSD symptoms which require specialised trauma treatment
* a suspected eating disorder defined as a BMI lower than 18,
* an IQ below 85,
* insufficient command of the Dutch language.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Generic sense of ability to adapt scale (GSAAS) | Up to 23 repeated measures, i.e. weekly over the course of 23 weeks (5-8 weeks control period + 10 weeks intervention + 5 weeks follow-up)
  Assessment of the ability to adapt with 10 5-point scale items.

SECONDARY OUTCOMES:
Self-expression and Emotion Regulation in Art Therapy Scale (SERATS) | Up to 23 repeated measures, i.e. weekly over the course of 23 weeks (5-8 weeks control period + 10 weeks intervention + 5 weeks follow-up)
  Self-expression and Emotion Regulation in Art Therapy Scale (SERATS): Assessment of emotional self-expression and regulation during therapy with 9 5-point scale items
Schema Modes Questionnaire, Healthy adult and Happy Child Subscale. (SMI) | Up to 23 repeated measures, i.e. weekly over the course of 23 weeks (5-8 weeks control period + 10 weeks intervention + 5 weeks follow-up)
  Assessment of adaptive schemamodes the Healthy adult and Happy Child, with 20 6-point scale items.
Schema Modes Questionnaire, maladaptive schemamodes. (SMI) | 2 repeated measures of the SMI the maladaptive modes, at the start of the control period and at the end of the follow up period, max. 23 weeks apart]
  Assessment of maladaptive schemamodes, with 98 6-point scale items.
Mental Health Continuum- short form (MHC-sf). | 2 repeated measures of the MHC-sf for Mental wellbeing, at the start of the control period and at the end of the follow up period, max. 23 weeks apart]
  Assessment of Mental wellbeing, with 14 6-point scale items
Brief Symptom Inventory (BSI). | 2 repeated measures of the BSI for, at the start of the control period and at the end of the follow up period, max. 23 weeks apart]
  Assessment of sympoms of psychopathology, with 53 5-points scale items.

OTHER OUTCOMES:
Interviews with the participants and therapists | Once 3 weeks after the intervention
  Semi structured interviews about the experiences of the participants and the therapists with the intervention, qualitative data.

CONTACTS AND LOCATIONS:
Overall Officials: Christine de Vries, MSc, Study Director — HAN University of Applied Sciences
Locations (1):
- HAN University of Applied Sciences, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make IPD available, but personal data will not be shared at all. Using a doi for the processed data giving a description of the meta-data and then data can be requested at the principal investigator, to whom data requests can be sent.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the main paper until 10 years after this publication.
Access Criteria: The principal investigator will investigate whether requests are reasonable and feasible and adhere to ethical considerations.

REFERENCES:
- [Background] Franken K, Schuffelen P, Ten Klooster P, van Doesum K, Westerhof G, Bohlmeijer E. Introduction of the generic sense of ability to adapt scale and validation in a sample of outpatient adults with mental health problems. Front Psychol. 2023 Mar 29;14:985408. doi: 10.3389/fpsyg.2023.985408. eCollection 2023. PMID 37063565
- [Background] Bohlmeijer E, Westerhof G. The Model for Sustainable Mental Health: Future Directions for Integrating Positive Psychology Into Mental Health Care. Front Psychol. 2021 Oct 21;12:747999. doi: 10.3389/fpsyg.2021.747999. eCollection 2021. PMID 34744925
- [Background] Franken, C.P.M., Vos, J.A. de, Westerhof, G.J., & Bohlmeijer, E. (2019). De Mental Health Continuum Short Form (MHC-SF), een handleiding voor behandelaren in de geestelijke gezondheidszorg voor het interpreteren en bespreken van scores met patiënten. Enschede; Universiteit Twente.
- [Derived] Wiersma IC, Wouters H, Timmerman K, Heijman J, Westerhof GJ, Radstaak M, Haeyen S. Promoting psychological adaptability and well-being of patients with personality disorders with creative arts and psychomotor therapies: protocol of an intervention mapping study. BMJ Open. 2024 Dec 31;14(12):e090275. doi: 10.1136/bmjopen-2024-090275. PMID 39740945